CLINICAL TRIAL: NCT02157337
Title: The Effect of Atorvastatin on Prevention of Postoperative Acute Kidney Injury in Patients Undergoing Aortic Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 4-2013-0551
Record Dates: First submitted 2014-06-03; First posted 2014-06-06 (Estimated); Last update posted 2017-01-25 (Estimated); Status verified 2017-01

CONDITIONS: Aortic Surgery; Acute Kidney Injury
Keywords: aortic surgery; postoperative acute kidney injury; statin; the patient undergoing aortic surgery
MeSH Terms: conditions — Acute Kidney Injury | interventions — Atorvastatin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- atrovastatin (Experimental)
  Interventions: Drug: Atorvastatin
- placebo (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Atorvastatin — 80 mg (PO) once daily for 6 days
  Arms: atrovastatin
Drug: placebo — 80 mg (PO) once daily for 6 days
  Arms: placebo

SUMMARY:
Acute kidney injury(AKI) is a common and severe complication after the cardiac surgery. Postoperative AKI increases the in-hospital stay, intensive care unit(ICU) stay and postoperative mortality. Aortic surgery is the most risky surgery that causes the postoperative AKI, and the incidence of AKI after aortic surgery is about 50%.

Statin is a 3-hydroxy-3-methyl-glutaryl co-enzyme A (HMG CoA) reductase inhibitors and is used primarily to lower the level of plasma cholesterol. Apart from the antilipid effect, statin has pleiotropic effects include anti-inflammation, decrease of oxidative stress, recovery of endothelial cell injury and stabilization of thrombus.

The pathology of AKI after aortic surgery include not only hypoperfusion of renal blood flow but also thromboembolism, inflammatory reaction after use of cardiopulmonary bypass(CPB) and oxidative stress. Therefore, the incidence of AKI after aortic surgery can be expected to decrease after the perioperative use of statin because of the pleiotropic effects of it. The aim of this study is to examine the association between preoperative statin treatment and the incidence of postoperative acute kidney injury(AKI) in patients undergoing aortic surgery

ELIGIBILITY:
Inclusion Criteria:

1. the patients undergoing aortic surgery
2. the age: 20~80 yrs

Exclusion Criteria:

1. taking the statin before the admission
2. having preoperative severe renal dysfunction (eGFR < 15 ml/min per 1.73 m2)
3. past history of liver disease OR serum AST/ALT increase > 2-fold from upper normal limit
4. past history of myopathy, myasthenia gravis, rhabdomyolysis OR increased creatinine kinase
5. drug or alcohol abuser
6. hypothyroidism
7. taking Macrolide, Azole antifungals, H2 antagonists, Cyclosporine, Omeprazole, Amiodarone, Fibrates and Niacin

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2014-03-12 (Actual); Primary Completion 2015-05-29 (Actual); Study Completion 2015-05-29 (Actual)

PRIMARY OUTCOMES:
Serum creatinine increase ≥0.3 mg/dl OR increase to 1.5-fold from baseline OR Urine output(U/O) < 0.5 ml/kg/h for 6 h | up to 7 days after the aortic surgery

SECONDARY OUTCOMES:
Serum creatinine increase >2.0-3.0-fold from baseline OR U/O < 0.5 ml/kg/h for 12 h | up to 7 days after the aortic surgery

OTHER OUTCOMES:
Serum creatinine increase >3.0-fold from baseline OR serum creatinine ≥4.0 mg/dl with an acute increase of at least 0.5 mg/dl OR U/O <0.3 ml/kg/h for 24 h OR anuria for 12 h OR need for RRT | up to 7 days after the aortic surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anesthesiology and Pain Medicine, Seoul, Seoul, South Korea